CLINICAL TRIAL: NCT06378307
Title: A Transferability Study on the Conditions for a Successful Inclusive Education
Acronym: TIAP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2022-06
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Inclusive Education
Keywords: inclusive education; disability; innovation; transferability; realist evaluation; complex intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students, families, professionals: Students with disabilities, students without disabilities, families, educational professionals, social workers and professionals/volunteers working in recreational activities

SUMMARY:
The investigators are conducting a realist evaluation study with a multi-case and qualitative design. The study aims to identify the conditions that promote successful students with disabilities inclusive education at school. This study is nested in the TIAP research (Research to explore the conditions transfer of innovations in the field of disability, with a view to developing a transfer framework).

DETAILED DESCRIPTION:
The TIAP study aims to study the transferability of a local innovation in the field of inclusive education in order to identify the functions that can be transferred. Grounded in a theory based evaluation (called realist evaluation) the TIAP study is a qualitative case study. The study population comprises various participant profiles including students with disabilities, students without disabilities, families, educational professionals, social workers and professionals/volunteers working in recreational activities. Participants will be recruited in two schools from a French department (Eure et Loir). In this department the intervention (also called innovation) is implemented. This intervention implies a complete transformation carried out by the service providers for students with intellectual deficiencies as well as the educational system. Students with disabilities go at school in their geographical area. They attend a standard classroom and have educational and therapeutical support offered by the local service provider (DAME : Dispositif d'Accompagnement Médico-Educatif ). Service providers are seen as ressources for education professionals.

Qualitative data will be collected by interviewers through individual or collective interviews, Data collection will be based on the configurational elements Contest, Mechanisms, Outcomes based on a realist evaluation.

ELIGIBILITY:
Inclusion Criteria:

Children with disabilities

* Under 15 years of age
* With a disability (notified by the Maison Départementale de l'Autonomie - MDA - for support by the local service provider (DAME : Dispositif d'Accompagnement Médico-Educatif)
* Enrolled in either the elementary school or middle school selected for the study
* Whose parents have not objected to their participation in the study

Children who do not have a disability

* Under 15 years of age
* In the same classroom as a student with a disability already participating in the study
* Whose parents did not object to their participation in the study

Families

* Father and/or mother, with parental authority, of a child with a disability participating in the study
* Over 18 years of age
* Not under guardianship or curatorship
* Have signed a study participation consent form

Education professionals:

* Working in one of the 2 schools selected for the study
* Working as (if possible, 1 representative from each of these professional categories):
* a member of the school's management team, the ULIS (Unité Unités Localisées pour l'Inclusion Scolaire) teacher, the teachers of the standard classroom of the disabled children taking part in the study.
* Members of the school life team (lunchtime, recess)
* professionals working towards inclusive education at the level of the school and the department
* Having signed a consent to participate in the study

Professionals of the service provider (DAME : Dispositif d'Accompagnement Médico-Educatif):

* Working in the service provider's sector of the school chosen for the research.
* Supporting a disabled child taking part in the research project
* Working within the DAME management team, i.e. a DAME specialist teacher, the DAME pedagogical coordinator, professionals providing different educational or therapeutic support (if possible, 1 representative from each of these professional categories).
* Having signed a consent form to participate in the study

Professionals who work with children during leisure time, outside school hours (if possible, 1 representative from each of these professional categories):

* Being professionals of associations of leisure centers, sports clubs ... and support a disabled child participating in the study
* Professionals working for the Espace Ressources Handicap, which coordinates these activities, and working in one of the 2 schools chosen for the study.
* Have signed a consent form to participate in the study

Exclusion Criteria: None for the different populations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children with and without disabilities, families and professionals
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of inclusive education on children with disabilities autonomy and social participation at school | Day 0
  Perceptions of students with disabilities on : learning practices and support, accessibility, inclusion climate in their school , peer relations at school.
Effect of inclusive education on children with disabilities autonomy and social participation in their proximal living environment (leisures participation) | Day 0
  Perceptions of students with disabilities during leisure participation on : support, accessibility, inclusion climate, peer relations in their living environment
Effect of inclusive education on social participation of families with children with disabilities | Day 0
  Perceptions of families on their social participation in their living environment